CLINICAL TRIAL: NCT03166917
Title: Shenzhen Hospital of Southern Medical University
Brief Title: Clinical Application of Personal Designed 3D Printing Implants in Bone Defect Restoration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: fang guofang (Other)
Responsible Party: Sponsor-Investigator, fang guofang, Shenzhen Hospital of Southern Medical University, Shenzhen Hospital of Southern Medical University
Organization: Shenzhen Hospital of Southern Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C1033429
Record Dates: First submitted 2017-05-24; First posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Defect; Internal Prosthetic Device, Implants and Grafts, Orthopedic, Bone Graft
MeSH Terms: interventions — Printing, Three-Dimensional

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printing implant (Experimental): 3D printing implant in bone defect
  Interventions: Procedure: 3D printing implant
- Autogenous bone grafting (Placebo Comparator): autogenous bone grafting in bone defect
  Interventions: Procedure: autogenous bone grafting

INTERVENTIONS:
Procedure: 3D printing implant — 3D printing implants in bone defect
  Arms: 3D printing implant
Procedure: autogenous bone grafting — 3D printing implants in bone defect
  Arms: Autogenous bone grafting

SUMMARY:
Objective: Clinical application of 3D printing implant in bone defect treatment.

Study design: multicenter randomized controlled study . Methods:patients randomly grouped according to register number into internal fixation and bone graft group and 3D printing group. Reconstruct 3D models ,evaluate models preoperatively , simulate surgery in computer,design 3D implant, and 3D print implants,perform surgery with 3D implants to achieve the greatest degree of physiological reconstruction.Evaluate surgical efficacy .

ELIGIBILITY:
Inclusion Criteria:

* Open fracture with bone defect
* Burst fracture of spine with bone defect
* Bone tumor with bone defect
* Bone tuberculosis with bone defect
* Nonunion with bone defect

Exclusion Criteria:

* Patients who can not tolerate anesthesia and surgery due to severe impairment of heart and lung function
* Systemic or local infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
operative time | 3 years

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - Zhujing hospital of southern medical university, Guanzhou
  - Shenzhen Hospital of Southern Medical University, Shenzhen

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Li X, Wang Y, Zhao Y, Liu J, Xiao S, Mao K. Multilevel 3D Printing Implant for Reconstructing Cervical Spine With Metastatic Papillary Thyroid Carcinoma. Spine (Phila Pa 1976). 2017 Nov 15;42(22):E1326-E1330. doi: 10.1097/BRS.0000000000002229. PMID 28498291
- [Background] Yang F, Chen C, Zhou Q, Gong Y, Li R, Li C, Klampfl F, Freund S, Wu X, Sun Y, Li X, Schmidt M, Ma D, Yu Y. Laser beam melting 3D printing of Ti6Al4V based porous structured dental implants: fabrication, biocompatibility analysis and photoelastic study. Sci Rep. 2017 Mar 28;7:45360. doi: 10.1038/srep45360. PMID 28350007
- [Background] Mustafa SF, Evans PL, Sugar AW, Key SJ. Streamlining the manufacture of custom titanium orbital plates with a stereolithographic three-dimensional printed model. Br J Oral Maxillofac Surg. 2017 Jun;55(5):546-547. doi: 10.1016/j.bjoms.2016.03.003. Epub 2017 Apr 6. No abstract available. PMID 28392025
- [Background] Tan XP, Tan YJ, Chow CSL, Tor SB, Yeong WY. Metallic powder-bed based 3D printing of cellular scaffolds for orthopaedic implants: A state-of-the-art review on manufacturing, topological design, mechanical properties and biocompatibility. Mater Sci Eng C Mater Biol Appl. 2017 Jul 1;76:1328-1343. doi: 10.1016/j.msec.2017.02.094. Epub 2017 Feb 24. PMID 28482501